CLINICAL TRIAL: NCT04058132
Title: Cerebrovascular Reactivity (CVR) Assessed With Functional Near Infrared Spectroscopy (fNIRS) as a Biomarker of Traumatic Cerebrovascular Injury (TCVI) Measured Longitudinally After Acute TBI in Military Personnel
Brief Title: Cerebrovascular Reactivity Assessed With fNIRS as a Biomarker of TCVI After Acute Traumatic Brain Injury in Military
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding ran out after unanticipated length of time ( for IRB approval, CRADA, and start letter
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kimbra Kenney, Service Chief, Research Operations, NICoE, WRNMMC & Professor, USUHS Service and Department: NICoE, WRNMMC & Neurology, USUHS, Uniformed Services University of the Health Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WRNMMC-2017-0048
Record Dates: First submitted 2019-08-07; First posted 2019-08-15 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic cerebrovascular injury; Functional Near Infrared Spectroscopy (fNIRS)
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Sildenafil Citrate; Carbon Dioxide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Exposures/interventions will be the same for healthy controls and participants with traumatic brain injury No blinding and no treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1: acute/subacute Traumatic Brain Injury (Other): Any gender, age 18-55 years who have had a traumatic brain injury within 30 days
  Interventions: Drug: Sildenafil Citrate 50Mg Tab; Device: functional Near-infrared Spectroscopy (fNIRS); Other: Carbon Dioxide (CO2) 5%; Other: Neuropsychological Assessments; Drug: Gadolinium contrast infusion; Procedure: Blood sample collection for research purposes; Other: Structural brain Magnetic Resonance Imaging (MRI
- Group 2: Non-TBI healthy control (HC) (Other): Any gender, age 18-55 years with no history of traumatic brain injury
  Interventions: Drug: Sildenafil Citrate 50Mg Tab; Device: functional Near-infrared Spectroscopy (fNIRS); Other: Carbon Dioxide (CO2) 5%; Other: Neuropsychological Assessments; Drug: Gadolinium contrast infusion; Procedure: Blood sample collection for research purposes; Other: Structural brain Magnetic Resonance Imaging (MRI

INTERVENTIONS:
Drug: Sildenafil Citrate 50Mg Tab — sildenafil citrate (Viagra®, Pfizer. Inc., NY, NY). Sildenafil citrate is designated chemically as 1-[[3-(6,7-dihydro-1-methyl-7-oxo-3-propyl-1Hpyrazolo[4,3-d]pyrimidin-5-yl)-4- ethoxyphenyl]sulfonyl]-4-methylpiperazine citrate. Sildenafil citrate is a white to off-white crystalline powder with a solubility of 3.5 mg/mL in water and a molecular weight of 666.7. For this study, we will use 50 mg tablets for the single dose studies.
  Other Names: Viagra®
Device: functional Near-infrared Spectroscopy (fNIRS) — Functional Near-Infrared Spectroscopy (fNIRS): Functional near-infrared spectroscopy (fNIRS) a noninvasive technique that can measure cerebrovascular reactivity (CVR) will be used to measure regional cerebral blood flow and cerebrovascular reactivity in the brain. The device (fNRIS100, fNIR Device LLC), uses laser emission diodes (730nm and 850nm)which in a headband that is worn on the front of the scalp and forehead. Surrounding detectors a few centimeters away detect the light as it scatters through the underlying tissues. The technique is able to detect changes in the absorption spectrum of the tissue corresponding to the concentrations of oxyhemoglobin (HbO2) and deoxyhemoglobin (HbR), and indicate local perfusion changes. fNIRS will be performed twice at each study visit, once before and once about 45 minutes after single dose administration of sildenafil 50 mg.
Other: Carbon Dioxide (CO2) 5% — Carbon Dioxide (CO2) 5% mixed with room air. Both the fNIRS procedure and one Magnetic Resonance Imaging (MRI) session at visits that include imaging will be done with a hypercapnia challenge for comparison.
  CO2 (hypercapnia) challenge is similar to holding one's breath. Participant will wear a nose clip and a mouth breathing apparatus while in the MRI scanner or sitting in a chair during the fNIRS procedure.
  During the 7-minute hypercapnia procedure, participants will breathe room air and then switch to room air mixed with 5% CO2, from one to the other for one minute each.
Other: Neuropsychological Assessments — TBI Neuropsychological Assessments: Study participants will be administered a set of Neuropsychological Tests designed by the NINDS Common Data Elements (CDEs) initiative for TBI, in order to provide a comprehensive and broad assessment of deficits commonly found after TBI. We anticipate that the neuropsychological battery will require approximately 1 hour to complete. The measures (pencil and paper exercises, questionnaires, and interview by the examiner) to be administered are: Glasgow Outcome Scale-Extended (GOS-E). Learning trials portion of the California Verbal Learning Test (CVLT-II): The Trail Making Tests A and B (TMT): Subsets of the Wechsler Adult Intelligence Scale (WAIS-IV) (Digit Symbol and Symbol Search): Behavioral Symptoms Inventory-18: Satisfaction with Life Scale (SWLS): Word Reading subtest of Wide Range Achievement Test (WRAT)-4: Rivermead Post-Concussion Symptom Questionnaire.
Drug: Gadolinium contrast infusion — Gadolinium contrast infusion: Brain MRI with gadolinium contrast: Dynamic contrast-enhanced (DCE) MRI with intravenous gadolinium-based contrast agents (GBCAs) to measure their transfer rate between intravascular and extravascular compartments as a marker of blood-brain barrier (BBB) permeability. For the DCE sequence, the participant is injected with the contrast agent through a heplock/iv in the scanner and the sequence takes about 15 min. Half-life of gadolinium is about 1 ½ hours and 90-98% clearance from the body in 24 hours in people with normal kidney function.
Procedure: Blood sample collection for research purposes — Serum and plasma (5 ml each) will be collected at at each study visit 10 m or 2 tsp. per visit or up to 40 ml or 8 tsp. over the 180 day course of the study). Samples will be collected by study personnel.
Other: Structural brain Magnetic Resonance Imaging (MRI — Structural brain Magnetic Resonance Imaging (MRI): The scanner used is a 3.0 Tesla MR (Model 750, General Electric Healthcare), which is equipped with a high-performance gradient subsystem and a 32-channel head coil (General Electric Healthcare). These scans involve lying still in a scanner for several minutes at a time which is tube shaped, using magnetism to take images of the brain. There is no radiation in MRI. The participants will have up to 3 research brain MRIs. Healthy controls will have 1 MRI session.
  Common TBI MRI techniques will be performed. Block-design BOLD fMRI during which there will be a 7 minute hypercapnia challenge will be done to assess brain blood flow and measure cerebral vascular reactivity (CVR).

SUMMARY:
The study includes people who have recently had a traumatic brain injury (TBI) and healthy controls who have not had a TBI and is designed to measure brain blood flow serially after a TBI. Studies have shown that small blood vessels in the brain may be injured during a TBI. The goal is to learn about brain blood vessel function from as early as the first week to 6 months after a TBI . The study uses Near Infrared Spectroscopy (NIRS) which uses small lights that detect oxygen levels in the blood, measuring blood flow in the brain. This is compared with magnetic resonance imaging (MRI). When blood flow increases in the brain in response to a stimulus, this is called cerebral vascular reactivity (CVR).

The study aims to learn about CVR using a few minutes of special breathing similar to breath holding while in an MRI (magnetic resonance imaging), and CVR measures after one dose of a common drug called sildenafil (generic Viagra) 50 mg taken once during CVR measurements at each of up to 4 visits. The investigators will measure CVR at different times during a 6-month period in participants who have had a TBI to see how CVR measures and blood vessels function during the first 6 months after a brain injury.

DETAILED DESCRIPTION:
Background and significance:

Currently, more that 5.3 million Americans (or 2% of the population) live with disabilities resulting from TBI. Among OEF/OIF Veterans, TBI incidence estimates as high as 23% have been reported, with mild TBI (mTBI) being the most common.1 This proposal addresses the recommendations of the consensus of scientific conferences by aiming to develop a biomarker of traumatic cerebrovascular injury (TCVI) which can be useful in clinical trials of therapies.

Substantial data point to traumatic cerebrovascular injury (TCVI) underlying a significant portion of TBI-related disability. 2 The cerebral vasculature is a highly plastic tissue making TCVI an attractive target for therapeutic intervention after TBI. Preliminary studies indicate that PDE5 inhibitors such as sildenafil (Viagra®) show promise as treatment for cerebrovascular dysfunction after TBI. 3,4

The investigators adapted MRI-Blood Oxygenation Level Dependent (BOLD) with hypercapnia challenge, to the portable, less expensive, office-based Near InfraRed Spectroscopy (NIRS) technology and incorporated hypercapnia challenge as the functional challenge with NIRS.

MRI- BOLD BOLD (with 5% carbon dioxide (CO2) hypercapnia challenge via the Douglas Bag method) and fNIRS (also with 5% CO2 hypercapnia challenge via the Douglas Bag method) in traumatic brain injury (TBI) and healthy controls. The complementary methods give similar results with a high degree of correlation in TBI patients compared to healthy controls. 5 Nitric Oxide (NO), the primary endogenous vasodilator in the brain, plays a prominent role. Specific PDE5 inhibitors have come into widespread use, the first is Sildenafil (Viagra®) for the treatment of erectile dysfunction and primary pulmonary hypertension. The beneficial effect of sildenafil is related to increased local CBF and enhanced neurogenesis, vasculogenesis, and axonal remodeling in the peri-infarct zone. 6-9 To date, there have been no longitudinal studies of CVR using functional NIRS from the acute to the subacute/chronic stages of TBI in humans.

Objectives of this study:

1. To measure over time brain blood flow using fNIRS (using lights on the scalp) with hypercapnia challenge (like breath holding for about a minute at a time) in 30 people who have had a brain injury, moderate and severe patients, and compare it to that of 10 age-matched uninjured controls, starting as early as within 29 days of injury with the goal of within 7 days and measuring each time at approximately 1, 3 and 6 months after injury to better understand the extent and timing of cerebrovascular reactivity (CVR) in the first 6 months after TBI.
2. To compare brain injury-related brain blood flow changes with clinical magnetic resonance imaging (MRI) and post-concussive symptoms measured by survey questionnaires, a neurologist's examination, testing to measure thinking ability, and learn about blood markers associated with traumatic brain injury.
3. To measure changes in CVR longitudinally before and after a single dose administration of a phosphodiesterase 5 inhibitor, sildenafil citrate, up to 4 study time points (first 29 days days and approximately 1, 3 and 6 months after TBI).
4. To compare CVR measurements by fNIRS versus BOLD MRI with hypercapnia challenge.
5. In conjunction with primary measurement of cerebrovascular reactivity using BOLD MRI, secondary measurement of cerebrovascular permeability will also be collected using DCE MRI.

Study Design The proposal is a 24-month project in which the investigators will conduct a prospective, longitudinal, observational study of up to 40 acute TBI patients and 10 healthy controls.

1. WRNMMC male and female military health care beneficiaries (active duty, veterans or DEERS eligible) aged 18 to 55 years, presenting with a diagnosis of moderate or severe (DoD criteria) traumatic brain injury (TBI) and healthy volunteers aged 18 to 55 years.
2. Study participants at WRNMMC will be recruited from eligible military healthcare beneficiaries presenting to the WRNMMC ED or admitted to WRNMMC for TBI within 1 week of injury (most through TBI inpatient consult service and likely on trauma surgery, neurosurgery, orthopedics, neurology, PMR and/or internal medicine inpatient services).

Procedures:

Participants will sign a consent form, attend scheduled visits, and be paid $50 for each blood sample collected from participants at each of the up to 4 visits over a 6 month period.

Participants will have an inverview about their injury and medical history and examination by a study physician, have a urine pregnancy test (if applicable), complete some questionnaires, have some memory and thinking tests, give a blood sample, and do some imaging.

Imaging Magnetic Resonance Imaging (MRI). One MRI before and after about 45 minutes of one dose of sildenafil 50mg. Each imaging session will use hypercapnia using a Douglas bag, equipped with a switch to allow rapid shifting every minute from room air to 5% CO2 mixed with room air over 7 minutes. This kind of imaging will be done at 2 or 3 of the visits. The 29-day visit is optional, so if the participant's first visit is at the 30-day visit they will have imaging at that visit and then again at the 6-month visit. No imaging at the 90-day visit.

* Also common TBI MRI techniques will be performed (e.g. high-resolution 3D T1-weighted, T2, T2*, diffusion tensor imaging, arterial spin labeling), as well as the following sequences:
* Dynamic contrast-enhanced (DCE) MRI with intravenous gadolinium-based contrast agents (GBCAs) Participant goes to Radiology and gets heplock, etc. (pregnancy test if female)

Structural MRI

Participant comes out of scanner to place oral piece/noseclip for MRI-BOLD c hypercapnia.

Quick T1 for co-registration, then MRI-BOLD c hypercapnia challenge (10-15 min) Participant comes out of the scanner and takes mouthpiece/nose clip off. Next,DCE sequence, the participant is injected with the contrast agent through a heplock/iv in the scanner and the sequence takes about 15 min.

TOTAL scanner time is approximately 75-90 min.

Functional near infrared spectroscopy (fNIRS) will be be performed twice at each study visit, once before and once about 45 minutes after single dose administration of sildenafil 50 mg.

Study Medication

The study medication is used to activate a change in brain blood flow during the observation and measurement of cerebrovascular reactivity.

The study drug will be sildenafil citrate (Viagra®, Pfizer. Inc.). For this study, the investigators will use 50 mg tablets for the single dose administration at each visit.

Collection of Human Biological Specimens

Serum and plasma (5 ml each) will be collected at at each study visit (10 ml per visit or up to 40 ml over the 180 day course of the study).

Length of participation in the study: Participants enrolled in the TBI Group will have up to four study visits over a period of approximately 6 months and be enrolled for that length of time. Non-TBI Control participants require only a single visit and will be discharged from the study after their study visit is complete and results have been recorded.

Risks and Discomforts

fNIRS with hypercapnia challenge

The investigators anticipate the following non-serious adverse events (likely, with event rate < 5%):

1. Slight discomfort from the NIRS band on the head
2. Minor warmth under the band from the light emitters after ~ 30 minutes of testing
3. Anxiety and/or panic attack during hypercapnia challenge
4. Headache during/after hypercapnia challenge.

However, there are well recognized adverse effects. The following lists the adverse events reported by at least 2% of patients taking sildenafil in flexible dose Phase 2/3 studies, and were more common at the 100 mg dose than at lower dose than this study will be using.

Adverse events attributed to sildenafil in placebo-controlled randomized trials Adverse Event % of patients on sildenafil reporting AE (n = 734) % of patients on placebo reporting AE (n = 725) Headache 16% 4% Flushing 10% 1% Dyspepsia 7% 2% Nasal Congestion 4% 2% Urinary Tract Infection 3% 2% Abnormal vision* 3% 0% Diarrhea 3% 1% Dizziness 2% 1% Rash 2% 1%

*Abnormal Vision: Mild and transient, predominantly color tinge to vision, but increased sensitivity to light or blurred vision. In these studies, only one patient discontinued due to abnormal vision.

Orthostatic hypotension is an infrequent adverse effect of sildenafil therapy. VIAGRA doses above 25 mg should not be taken within 4 hours of taking an alpha-blocker.

Study participants will also be given the contact information for one of the study investigator physicians.

Neurocognitive tests Testing is critical for studying the effect of TBI on memory, behavior and functioning. All testing will be performed by a trained research assistant or psychometrist. No serious adverse events are anticipated.

Boredom Fatigue Frustration

Phlebotomy

Trained study personnel will draw 10 ml (2 teaspoons) at each study visit. Possible non-serious adverse events:

Bleeding Bruising Infection

Magnetic Resonance Imaging:

MRI has been safely performed in millions of persons; research subjects will be screened for metallic foreign bodies or other contraindications, similar to all clinical patients. Pregnant females will also be excluded from participating in these research MRIs.

Subjects may experience discomfort or anxiety while lying in the magnet and may communicate with the MRI technologist. Participants will have hearing protection.

Gadolinium-Based Contrast Agents:

Risks include local side effects from IV placement and contrast injection, systemic reaction to the MR contrast agents (less common than with CT contrast agents), and a rare but serious disease called nephrogenic systemic fibrosis (NSF).

There have been more recent descriptions of gadolinium deposition in the brain after exposure to MR contrast agents. The clinical significance (if any) of this discovery is currently unknown.

Subject Withdrawal

As stated in the consents, and as will be explained to the subjects, subjects may withdraw their participation from the study, at any time, without explanation. The procedure for withdrawal is stated in the consent document.

Privacy

All screening and enrollment procedures will be conducted in the study site clinics. All recruitment and subsequent study-related activities involving face-to-face interactions with subjects will be conducted in a private, closed-door office setting. All telephone contacts will be carried out in a closed room.

Confidentiality Protection

Each subject will be assigned a numerical code for identification purposes pertaining to data and biospecimens. The numberical code will contain no identifiers (numerical code only). A computer file linking subjects to their assigned numerical code will be safely stored as an encrypted file on a password protected computer. Paper records will be stored in locked cabinets in locked office space. Linking files will be kept for the life of the study and then destroyed. No subject will be identified in future publications as having taken part in this study.

ELIGIBILITY:
Inclusion Criteria (See Table 2 for more details)

1. Age 18 to 55 years, inclusive
2. Either gender
3. TBI subjects ONLY: Meets DoD criteria for moderate or severe TBI and TBI occurred less than 30 days prior to study enrollment (Sustained a traumatically induced physiological disruption of brain function, as manifested by at least one of the following:

   1. . Period of loss of consciousness > 30 minutes
   2. . Loss of memory for events lasting> 24 hours after the accident
   3. . Alteration of mental state lasting> 24 hours after the accident (e.g., feeling dazed, disoriented, and confused)
   4. . Clinical neuroimaging intracranial abnormality.

      * Traumatically induced includes the head being struck, the head striking an object, or the brain undergoing an acceleration/deceleration movement (i.e. whiplash) without direct external trauma to the head.
4. Ability to undergo fNIRS testing with hypercapnia challenge serially
5. Ability to provide informed consent.

Exclusion Criteria:

1. Unstable respiratory or hemodynamic status
2. Evidence of penetrating brain injury
3. TBI requiring craniotomy or craniectomy
4. History of disabling pre-existing neurologic disorder, e.g. dementia, uncontrolled epilepsy, multiple sclerosis, strokes, brain tumors, prior severe TBI, or other disorder that confounds interpretation of NIRS testing or neuropsychological results
5. History of pre-existing disabling mental illness, e.g. major depression or schizophrenia
6. Exclusion criteria for sildenafil:

   History of melanoma; Current use of organic nitrate vasodilators; Use of ritonavir (HIV-protease inhibitor); Current use of erythromycin, ketoconazole, or itraconazole; Current use of cimetidine; Current use of Alpha-blockers such as doxazosin (Cardura), tamsulosin (Flomax), and terazosin (Hytrin) prazosin (Minipress); Resting hypotension (systolic BP <90); Severe renal insufficiency; Hepatic cirrhosis; Cardiac failure or coronary artery disease causing unstable angina; Retinitis pigmentosa; Pregnant or breastfeeding female; Known hypersensitivity or allergy to sildenafil.
7. Inability to read and communicate in English
8. Exclusion criterion for healthy subjects only: History of TBI.
9. Current use of a PDE5 inhibitor (a drug such as Sildenafil, Tadalafil, Vardenafil, Avanafil, Udenafil,Dipyridamole, Vardenafil hydrochloride)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Detection of variation of oxyhemoglobin and deoxyhemoglobin concentration using a power analysis between groups during the hypercapnia challenge pre and post a single dose of sildenafil 50 mg at the specified time points after a TBI. | 2 years
  This is a pilot study, whose primary aim is to obtain pilot data that can be used to design a carefullypowered Phase III clinical trial. Thus, a power analysis is only an approximation.This compares favorably with the effect size of 1.3 noted in our preliminary study in chronic TBI (Figs. 2 and 4). For the observed effect size of 1.3, power will be 90%. Since we anticipate that the reduction in CVR will be greater in the acute period than in the chronic period, the proposed study has adequate sample size to measure the evolution of CVR over the subacute period after TBI. Sample size was calculated using GraphPad StatMate, v. 2.0 for Windows (GraphPad Software, San Diego, CA). The following assumptions were made: alpha =0.05, delta = 0.44, sigma = 0.40.
Longitudinal measure of CVR between groups | 2 years
  For each TBI, we will perform a one way ANOVA test between CVR measure for all the source/detectors pair at the different time point. At each time point of the study, we will also perform a t test on the mean CVR between the TBI group and the HC group.

CONTACTS AND LOCATIONS:
Overall Officials: Kimbra Kenney, MD, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
none collected

REFERENCES:
- [Result] Hoge CW, McGurk D, Thomas JL, Cox AL, Engel CC, Castro CA. Mild traumatic brain injury in U.S. Soldiers returning from Iraq. N Engl J Med. 2008 Jan 31;358(5):453-63. doi: 10.1056/NEJMoa072972. Epub 2008 Jan 30. PMID 18234750
- [Result] Washington CW, Derdeyn CP, Dhar R, Arias EJ, Chicoine MR, Cross DT, Dacey RG Jr, Han BH, Moran CJ, Rich KM, Vellimana AK, Zipfel GJ. A Phase I proof-of-concept and safety trial of sildenafil to treat cerebral vasospasm following subarachnoid hemorrhage. J Neurosurg. 2016 Feb;124(2):318-27. doi: 10.3171/2015.2.JNS142752. Epub 2015 Aug 28. PMID 26314998
- [Result] Nicolakakis N, Aboulkassim T, Aliaga A, Tong XK, Rosa-Neto P, Hamel E. Intact memory in TGF-beta1 transgenic mice featuring chronic cerebrovascular deficit: recovery with pioglitazone. J Cereb Blood Flow Metab. 2011 Jan;31(1):200-11. doi: 10.1038/jcbfm.2010.78. Epub 2010 Jun 23. PMID 20571524
- [Result] Nicolakakis N, Hamel E. Neurovascular function in Alzheimer's disease patients and experimental models. J Cereb Blood Flow Metab. 2011 Jun;31(6):1354-70. doi: 10.1038/jcbfm.2011.43. Epub 2011 Apr 6. PMID 21468088
- [Result] Amyot F, Kenney K, Moore C, Haber M, Turtzo LC, Shenouda C, Silverman E, Gong Y, Qu BX, Harburg L, Lu HY, Wassermann EM, Diaz-Arrastia R. Imaging of Cerebrovascular Function in Chronic Traumatic Brain Injury. J Neurotrauma. 2018 May 15;35(10):1116-1123. doi: 10.1089/neu.2017.5114. Epub 2018 Mar 20. PMID 29065769
- [Result] Zhang R, Wang Y, Zhang L, Zhang Z, Tsang W, Lu M, Zhang L, Chopp M. Sildenafil (Viagra) induces neurogenesis and promotes functional recovery after stroke in rats. Stroke. 2002 Nov;33(11):2675-80. doi: 10.1161/01.str.0000034399.95249.59. PMID 12411660
- [Result] Li L, Jiang Q, Zhang L, Ding G, Gang Zhang Z, Li Q, Ewing JR, Lu M, Panda S, Ledbetter KA, Whitton PA, Chopp M. Angiogenesis and improved cerebral blood flow in the ischemic boundary area detected by MRI after administration of sildenafil to rats with embolic stroke. Brain Res. 2007 Feb 9;1132(1):185-92. doi: 10.1016/j.brainres.2006.10.098. Epub 2006 Dec 26. PMID 17188664
- [Result] Ding G, Jiang Q, Li L, Zhang L, Zhang ZG, Ledbetter KA, Panda S, Davarani SP, Athiraman H, Li Q, Ewing JR, Chopp M. Magnetic resonance imaging investigation of axonal remodeling and angiogenesis after embolic stroke in sildenafil-treated rats. J Cereb Blood Flow Metab. 2008 Aug;28(8):1440-8. doi: 10.1038/jcbfm.2008.33. Epub 2008 Apr 16. PMID 18418368
- [Result] Atalay B, Caner H, Cekinmez M, Ozen O, Celasun B, Altinors N. Systemic administration of phosphodiesterase V inhibitor, sildenafil citrate, for attenuation of cerebral vasospasm after experimental subarachnoid hemorrhage. Neurosurgery. 2006 Nov;59(5):1102-7; discussion 1107-8. doi: 10.1227/01.NEU.0000245605.22817.44. PMID 17143244